CLINICAL TRIAL: NCT05668793
Title: Methylation Detection of KCNA3 and OTOP2 Genes in Plasma for the Auxiliary Diagnosis of Hepatocellular Carcinoma: a Clinical Trial
Brief Title: GNB4 and Riplet Gene Methylation Combined Detection Kit (Fluorescence PCR Method)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Wuhan Ammunition Life-tech Co., Ltd (Industry)
Collaborators: Wuhan University (Other)
Responsible Party: Sponsor
Other Study IDs: AD07
Record Dates: First submitted 2022-12-09; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma diagnosis; methylation; GNB4; Riplet; Fluorescence PCR
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — 1. Sample type: Human plasma samples.
  2. Sample collection: Choose a blood collection vessel containing EDTA anticoagulant for blood collection, and gently turn it upside down after blood collection.
     Repeat 8-10 times and mix gently.The blood collection volume is not less than 10 mL.
  3. Sample preservation:The collected blood samples should be centrifuged immediately to prepare plasma. If they cannot be processed in time, they should be stored at room temperature (15℃~30℃) for no more than 3 hours, or at 2℃~8℃ for no more than 8 hours, and whole blood should not be frozen.
  Plasma samples can be stored at 2℃~8℃ for no more than 18 hours, at -25℃~-15℃ for no more than 28 days, and at -80℃±5℃ for no more than 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive group: The positive group is composed of patients with hepatocellular carcinoma of different stages and pathological types.
  Interventions: Diagnostic Test: GNB4 and Riplet Gene Methylation Combined Detection Kit (Fluorescent PCR Method)
- Negative group: 1. Patients with other digestive system malignancies (including stomach cancer, esophageal cancer, colorectal cancer, pancreatic cancer, gallbladder/duct cancer, etc.), patients with non-digestive system malignancies (including lung cancer, thyroid cancer, cervical cancer, endometrial cancer, breast cancer, prostate cancer, urothelial cancer, etc.).
  2. Patients with benign liver diseases (such as cirrhosis, hepatitis, fatty liver, liver adenoma, liver cyst, etc.).
  Interventions: Diagnostic Test: GNB4 and Riplet Gene Methylation Combined Detection Kit (Fluorescent PCR Method)

INTERVENTIONS:
Diagnostic Test: GNB4 and Riplet Gene Methylation Combined Detection Kit (Fluorescent PCR Method) — Blood samples from participants in the group were collected and methylation tests were performed according to the kit instructions.

SUMMARY:
The goal of this observational study is to test the clinical efficacy of "GNB4 and Riplet gene methylation combined detection kit (fluorescence PCR method)"in hepatocellular carcinoma auxiliary diagnosis. The main questions it aims to answer are:

1. How consistent are the test results of the kit with the clinical reference diagnostic criteria?
2. Sanger sequencing can visually show whether each sample contains methylation sites, so in this clinical trial, the kit results were compared with Sanger sequencing results to analyze the reagent's accuracy in detecting GNB4 and Riplet gene methylation.

Each participant is required to provide no less than 10 ml of blood to complete the kit test.

DETAILED DESCRIPTION:
1. Before the start of clinical trials, investigators will be uniformly trained by experts from the clinical trial institutions or from the sponsor. Researchers should be familiar with and correctly operated the test kits and instruments.
2. Throughout the clinical trial process, the clinical trial institution should ensure that it follows the scheduled protocal and strictly abide by the instructions of instruments and reagents.
3. The entire trial process should be completed by the researchers in the laboratory of the clinical trial institution. Except for the necessary guidance, the technical staff of the sponsor shall not interfere with the experimental process at will, especially data collection process. Blind methods should be used to ensure the objectivity of the test results.
4. The sponsor shall ensure that the test reagents are qualified, and transported to the clinical institution in accordance with the transportation conditions in the manual. Researchers should record the information of receipt, storage, use, handling and recycling process.
5. Researchers should ensure that the clinical trial data are recorded accurately, completely, clearly and in a timely manner. Any changes to the data should be signed and dated by the researcher, and the original records should be kept. The original records should be clear and recognizable. All observations and findings in clinical trials should be truthfully recorded and verified to ensure the reliability of the data and to ensure that the conclusions of clinical trials are derived from the original records.

ELIGIBILITY:
Inclusion Criteria:

* Those who meet any of the following conditions can be enrolled into the hepatocellular carcinoma group：

  1. Patients who have suspected placeholder lesions in the liver area after existing examinations and plan to undergo multi-parameter MRI, CT dynamic enhancement scans, ultrasound imaging or enhanced magnetic resonance scans with the hepatocyte-specific contrast agent disodium gadolinium cerate (Gd-EOB-DTPA)；
  2. Patients who are highly suspected of liver cancer diagnosed by multi-parameter MRI, CT dynamic enhancement scan, ultrasound contrast, liver cell-specific contrast agent disodium gadolinium cerate (Gd-EOB-DTPA) enhanced magnetic resonance scan or puncture biopsy, before treatment and surgery；
* Those who meet any of the following conditions can be enrolled into the negative group：

  1. Patients with benign liver diseases (including cirrhosis, hepatitis, fatty liver, liver adenoma, liver cyst, etc.).
  2. Untreated patients with other digestive system tumors (including stomach cancer, colorectal cancer, esophageal cancer, pancreatic cancer, gallbladder/duct cancer, etc.) and patients with non-digestive system tumors (including lung cancer, thyroid cancer, cervical cancer, endometrial cancer, breast cancer, prostate cancer, urothelial cancer, etc.).

Exclusion Criteria:

Those who meet any of the following conditions should be excluded：

1. Patients with hepatocellular carcinoma who have received anti-tumor treatments such as radiotherapy/chemotherapy；
2. Hepatocellular carcinoma patients suffering from other malignant tumors at the same time；
3. Samples that are not kept as required or samples of hemolysis；
4. The sample size collected does not meet the testing requirements；

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. The number of patients with hepatocellular carcinoma should be not less than 350, and should cover different stages and different pathological types.
  2. The number of patients with other malignancies of the digestive system should not be less than 200.
  3. The number of patients with benign liver disease should not be less than 300.
  4. The number of all samples enrolled should be not less than 1000 cases.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
validity | immediately after the procedure
  In this study, validity indicates the consistency of methylation test with the clinical reference diagnostic standards, including sensitivity and specificity. Sensitivity indicates the proportion of methylation-positive samples in hepatocellular carcinoma samples. Specificity indicates the proportion of methylation-negative samples in nagative group.

SECONDARY OUTCOMES:
reliability | immediately after the procedure
  In this study, the reliability evaluation included two indicators, namely the agreement rate of methylation detection with Sanger sequencing, and the Kappa value of the two methods.

IPD SHARING:
Plan to Share IPD: No
Confidential information of the individual participant will be retained by investigators and clinical trial institutions, any personal information of subjects will not be disclosed in reports, publications, etc.
  Direct access to source data and and files is only allowed for the purpose of monitoring, auditing or inspection, without revealing the subject's privacy.
  The medical products administration may inspect the basic documents of clinical trials of medical devices in order to confirm the authenticity and the integrity of the collected data.